CLINICAL TRIAL: NCT04504201
Title: Clinic-based "Patient-Centered Communication About Healthy Weight" (PCC-HW) in a Diverse Sample of Women With Early Breast Cancer
Brief Title: Patient-centered Communication About Healthy Weight in Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: LCCC 1954
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Breast Cancer Patients: Early breast cancer patients (Stage I-III) who have completed primary treatment with a current Body mass index (BMI) over 30.
  Interventions: Other: Focus Group
- Medical Oncology Clinicians: Oncology providers associated with community-based practices
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Focus Group — Breast cancer patients and oncology clinicians will participate in separate focus groups discussing patient-centered communication about healthy weight.

SUMMARY:
Comorbidities in breast cancer survival account for 49% of overall survival difference between black and white women. Many obesity-related comorbidities disproportionately affect black women, therefore pointing to a need to address obesity related comorbidities in survival disparities in early breast cancer patients. This study tinvestigates how messages and messaging about healthy weight can be tailored for racially diverse breast cancer survivors with obesity in order to ensure that clinic-based communications between patients and their oncology provider are patient-centered and culturally sensitive.

DETAILED DESCRIPTION:
The overall goal of this research is to collect essential input for the future development of a quality improvement intervention to foster "Patient-Center Communication about Healthy Weigh in clinical practice

Primary Objective:

1. Understand patient-centered perspectives on health weight communication with oncology clinicians by conducting focus groups

   Secondary Objective
2. Understand oncology clinician perspectives on patient center communications for healthy weight interactions through semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria for Breast Cancer Cohort:

* Age 21 or older
* Diagnosed with early breast cancer, Stages I-III
* Completed primary treatment (Surgery, chemotherapy, radiation) within past 2 years
* Body mass Index of equal or greater than 30

Exclusion Criteria:

* Cannot understand and speak English

INclusion Criteria for Oncology provider cohort:

* Breast cancer oncology provider in North Carolina with MD/DO/PA/NP/RN
* associated with community-based practices

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer patients and Breast oncology providers will be eligible for this study
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Feedback from patients regarding healthy weight communication through focus groups | 3 year
  Summary of conversation based on 5A's Behavioral Change Model

SECONDARY OUTCOMES:
Feedback from oncology providers regarding healthy weight communication through semi-structured interview | 3 year
  Provider suggestions on how to implement 5A's Behavioral change model into patient care

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nyrop, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States